CLINICAL TRIAL: NCT07313982
Title: RILEVANZA DIAGNOSTICA DELLA ESPRESSIONE DI LEF-1 NEL LINFOMA A PICCOLI LINFOCITI/LEUCEMIA LINFATICA CRONICA B
Brief Title: LEF1 EXPRESSION IN B-CELL CHRONIC LYMPHOCYTIC LEUKEMIA PATIENTS: A MARKER FOR DIAGNOSIS AND SURVIVAL PREDICTION
Acronym: LLC/LEF1 2024
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Elena Sabattini, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: LLC/LEF1 2024
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Tissue. Formalin-fixed, paraffin-embedded samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic lymphocytic leukemia (CLL) is a highly heterogeneous B-cell hematological malignancy characterized by clonal expansion and accumulation of morphologically mature B-lymphocytes with a peculiar immunophenotype in peripheral blood, bone marrow, and secondary lymphoid tissues. Diagnosis is usually possible by flow cytometry, while lymph node and/or bone marrow biopsy may be helpful if immunophenotyping is inconclusive. A better understanding of pathogenesis has, recently, allowed the identification of new markers, improving patient stratification, implementing the therapeutic armamentarium with new agents targeting key intracellular signaling pathways. The canonical Wnt/β-catenin pathway is well recognized and known to drive malignant transformation of several cancer types including B-CLL. High expression of WNT3 and its transcription factor LEF1 in CLL considered as one of the strongest facts supporting the role of this pathway in CLL.

The evaluation of LEF-1 expression by immunohistochemistry in the diagnostic setting is still limited and a substantial number of CLL patients with negative LEF-1 expression has been reported. This is a study of LEF-1 expression to test the utility of using it for optimizing the B-CLL diagnosis and correlate it with the immunohistochemical, clinical and molecular data and compare LEF-1 negative and positive cases to identify a possible LEF-1 expression related signature that could be useful in differential diagnosis, in prognostic stratification and possibility of using targeted drugs

DETAILED DESCRIPTION:
Small lymphocytic lymphoma/chronic lymphocytic leukemia (SLL/CLL) is the most common chronic leukemia in adults in Western countries. SLL/CLL is classified as a chronic lymphoproliferative disorder within the category of mature B-cell neoplasms according to the World Health Organization (WHO) classification, and is characterized by the relentless accumulation of mature B lymphocytes displaying a distinctive immunophenotype. The disease may involve peripheral blood, bone marrow, lymph nodes, and the spleen. The median age at diagnosis is approximately 70 years, although about 10% of cases occur in young adults, and males are affected more frequently than females. In Western countries, the incidence is 2-6 cases per 100,000 inhabitants per year, increasing with age.¹ The clinical course of CLL is highly heterogeneous: most patients have an indolent course requiring no therapy or delayed treatment with prolonged survival, whereas others present with an aggressive disease requiring early treatment and experiencing frequent relapses.

SLL/CLL is generally diagnosed during routine blood testing in asymptomatic patients who exhibit absolute lymphocytosis, often with Gumprecht shadows visible on peripheral blood smears (representing fragile lymphocytes disrupted during slide preparation). The diagnosis of SLL/CLL is based on the presence of ≥5,000/µl clonal B lymphocytes in peripheral blood, which on flow cytometry are CD19+, CD5+, CD23+, CD200+, with dim CD20 expression, weak CD22 and/or CD79b, and weak surface immunoglobulin expression with light-chain restriction. Diagnosis is usually achievable through immunophenotyping of peripheral blood, whereas lymph node biopsy and/or bone marrow biopsy may be useful when immunophenotyping is inconclusive.

In the diagnostic work-up of SLL/CLL, CD5, CD19, CD20, CD23, and surface or cytoplasmic kappa/lambda light chains are considered essential markers, while CD10, CD43, CD79b, CD81, CD200, and ROR1 serve as additional antigens useful for differential diagnosis among small B-cell lymphomas/leukemias. Beyond assessing del(11q), del(13q), del(17p), and trisomy 12, TP53 mutational analysis and evaluation of somatic hypermutation (SHM) of the immunoglobulin heavy-chain variable region (IGHV) are essential for comprehensive prognostic assessment in SLL/CLL. IGHV mutational status and TP53 status are included in the CLL International Prognostic Index (CLL-IPI), together with age, clinical stage, and β2-microglobulin levels. Assessment of karyotypic complexity and the mutational status of BTK, PLCG2, and BCL2 remain desirable additional investigations within a targeted-therapy approach.

In recent years, improved understanding of SLL/CLL pathogenesis has clarified preneoplastic conditions (e.g., monoclonal B-cell lymphocytosis), enabled identification of novel diagnostic, prognostic, and predictive markers, refined patient stratification, and expanded the therapeutic armamentarium with new agents targeting key intracellular signaling pathways. Among these, several studies have demonstrated dysregulation of the WNT/β-catenin pathway in SLL/CLL. The final mediator of this pathway is LEF-1 (lymphoid enhancer-binding factor 1), a key transcription factor regulating cell proliferation and survival and playing a fundamental role in lymphopoiesis. LEF-1 is normally expressed in a subset of T cells and in B-cell precursors but is silenced in mature B cells; however, gene expression profiling studies have shown overexpression of LEF-1 in SLL/CLL compared with normal B cells. This expression is detectable by immunohistochemistry in tissue samples, where its presence has been confirmed. Nonetheless, although LEF-1 expression has demonstrated usefulness in distinguishing SLL/CLL from other indolent B-cell lymphomas, its diagnostic application remains limited. Moreover, a subset of CLL patients does not express LEF-1, and the characteristics of these patients have not yet been investigated.

The aim of this study, with an anticipated enrollment of up to 350 patients with a confirmed diagnosis of SLL/CLL and available molecular data at diagnosis, is to re-evaluate immunohistochemical expression on biopsy specimens (most commonly bone-marrow biopsies) to:

1. confirm actual LEF-1 expression positivity, and
2. statistically assess potential clinical correlations between LEF-1-positive and LEF-1-negative subsets, in an effort to identify possible diagnostic, prognostic, or therapeutic implications.

The study is observational, multicenter, national, retrospective/ Prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of SLL/CLL - B
* Males and females, adults at diagnosis
* Patients with available tissue (lymph node, extralymph node, or bone marrow) on which immunohistochemical analysis including LEF-1 has been performed and who have already submitted mutational and/or cytogenetic analysis data.

Exclusion Criteria:

* - Patients with LEF1-positive indolent B-cell lymphomas not supported by a genetic evaluation with SSL/CLL.
* CLL cases for which a biopsy is not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with SLL/CLL who turned to the Hemolymphatic Pathology Unit of the IRCCS - Bologna University Hospital, Policlinico S. Orsola-Malpighi, and the Hemolymphatic Pathology Unit of the Pathological Anatomy Unit, Policlinico Universitario Umberto I, Rome, from January 2014 to December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
LEF1 expression | From the beginning of the study to the analysis of all the results: 24 months
  To evaluate the expression of the LEF-1 molecule at diagnosis, in a cohort of patients with a clinical and histopathological diagnosis of SLL/CLL, with an expected value of around 70% of positive cases.

SECONDARY OUTCOMES:
Relationship | From the beginning of the study to the analysis of all the results: 24 months
  To evaluate the relationship between immunohistochemical and mutational parameters collected at diagnosis and clinical data.
New markers | From the beginning of the study to the analysis of all the results: 24 months
  Identify new possible diagnostic, prognostic or therapeutic markers.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Azienda Ospedaliero-Universitaria Di Bologna, Bologna, BOLOGNA, Italy